CLINICAL TRIAL: NCT06941727
Title: Association Between Maximum Mouth Opening and Masseter Muscle Elasticity in Oral Cancer Patients: A Study Using Sonographic Elastography
Brief Title: Relationship Between Mouth Opening and Masseter Elasticity in Oral Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202502031RIN
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-02

CONDITIONS: Oral Cancer
Keywords: Maximum interincisal opening; Elastography; Masseter muscle; Elasticity
MeSH Terms: conditions — Mouth Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: ultrasonographic imaging — masseter muscle elasticity

SUMMARY:
The study aims to assess the hardness of masticatory muscles in post-surgical oral cancer patients using strain elastography ultrasound, calculating the masseter elasticity index and exploring its association with maximum interincisal mouth opening. Furthermore, the study incorporates exercise training to analyze whether changes in masseter hardness can serve as an objective indicator for predicting the improvement of trismus.

DETAILED DESCRIPTION:
This study aims to evaluate the hardness of masticatory muscles in patients who have undergone surgery for oral cancer, using strain elastography ultrasound. Specifically, the research focuses on measuring the elasticity of the masseter muscle by calculating the masseter elasticity index (MEI) and analyzing its correlation with maximum interincisal mouth opening (MIO). Since trismus, or restricted mouth opening, is a common post-surgical complication affecting oral function and quality of life, understanding the relationship between muscle elasticity and jaw mobility is crucial. Additionally, the study incorporates a structured exercise training program designed to improve jaw function in these patients. By monitoring changes in masseter muscle hardness before and after the intervention, the research aims to determine whether variations in muscle elasticity can serve as an objective indicator for predicting improvements in trismus.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed oral cancer patients who are scheduled to receive cancer-related treatments (e.g., oral cancer surgery, radiotherapy, chemotherapy, or chemoradiotherapy).
2. Age between 20 and 65 years.

Exclusion Criteria:

1. Could not communicate.
2. Had any disorder that could influence movement performance.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 10 patients, aged 20 to 65 years, are first diagnosed with oral cancer and underwent surgery and routine physical therapy within three months.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Masseter muscle elasticity | Pre-intervention, 8 weeks post-intervention
  The masseter elasticity index is calculated as the ratio of the average elasticity of the masseter muscle to that of the isolation-coupling Pad (icPad).
Maximum interincisal mouth opening | Pre-intervention, 8 weeks post-intervention
  Maximum interincisal mouth opening is measured using a mouth-opening ruler, placed at the edges of the upper and lower central incisors to determine the distance.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, Principal Investigator — National Taiwan University, College of Medicine

REFERENCES:
- [Background] Yeh SA, Tang Y, Lui CC, Huang YJ, Huang EY. Treatment outcomes and late complications of 849 patients with nasopharyngeal carcinoma treated with radiotherapy alone. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):672-9. doi: 10.1016/j.ijrobp.2004.11.002. PMID 15936544
- [Background] Taljanovic MS, Gimber LH, Becker GW, Latt LD, Klauser AS, Melville DM, Gao L, Witte RS. Shear-Wave Elastography: Basic Physics and Musculoskeletal Applications. Radiographics. 2017 May-Jun;37(3):855-870. doi: 10.1148/rg.2017160116. PMID 28493799
- [Background] Takashima M, Arai Y, Kawamura A, Hayashi T, Takagi R. Quantitative evaluation of masseter muscle stiffness in patients with temporomandibular disorders using shear wave elastography. J Prosthodont Res. 2017 Oct;61(4):432-438. doi: 10.1016/j.jpor.2017.01.003. Epub 2017 Feb 7. PMID 28188109
- [Background] Karlsson O, Karlsson T, Pauli N, Andrell P, Finizia C. Jaw exercise therapy for the treatment of trismus in head and neck Cancer: a prospective three-year follow-up study. Support Care Cancer. 2021 Jul;29(7):3793-3800. doi: 10.1007/s00520-020-05517-7. Epub 2020 Nov 24. PMID 32435968
- [Background] Itoh A, Ueno E, Tohno E, Kamma H, Takahashi H, Shiina T, Yamakawa M, Matsumura T. Breast disease: clinical application of US elastography for diagnosis. Radiology. 2006 May;239(2):341-50. doi: 10.1148/radiol.2391041676. Epub 2006 Feb 16. PMID 16484352
- [Background] Chen YH, Liang WA, Hsu CY, Guo SL, Lien SH, Tseng HJ, Chao YH. Functional outcomes and quality of life after a 6-month early intervention program for oral cancer survivors: a single-arm clinical trial. PeerJ. 2018 Feb 21;6:e4419. doi: 10.7717/peerj.4419. eCollection 2018. PMID 29492348
- [Background] Cardoso RC, Kamal M, Zaveri J, Chambers MS, Gunn GB, Fuller CD, Lai SY, Mott FE, McMillan H, Hutcheson KA. Self-Reported Trismus: prevalence, severity and impact on quality of life in oropharyngeal cancer survivorship: a cross-sectional survey report from a comprehensive cancer center. Support Care Cancer. 2021 Apr;29(4):1825-1835. doi: 10.1007/s00520-020-05630-7. Epub 2020 Aug 11. PMID 32779007
- [Background] Ariji Y, Nakayama M, Nishiyama W, Nozawa M, Ariji E. Shear-wave sonoelastography for assessing masseter muscle hardness in comparison with strain sonoelastography: study with phantoms and healthy volunteers. Dentomaxillofac Radiol. 2016;45(2):20150251. doi: 10.1259/dmfr.20150251. Epub 2015 Dec 1. PMID 26624000